CLINICAL TRIAL: NCT00350051
Title: Phase 2 Study of ZK-Epothilone (ZK-Epo; ZK219477) Plus Prednisone as First-line Chemotherapy in Patients With Metastatic Androgen-independent Prostate Cancer
Brief Title: ZK-Epo Given With Prednisone in Patients With Metastatic Androgen-independent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91500; 307976 (Other: Company internal); NCT00430222 (obsolete NCT alias)
Record Dates: First submitted 2006-07-07; First posted 2006-07-10 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Metastatic androgen-independent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sagopilone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Sagopilone (ZK 219477) + prednisone

INTERVENTIONS:
Drug: Sagopilone (ZK 219477) + prednisone — Chemotherapy for hormone refractory prostate cancer; 16mg/m2 (up to 32mg/m2 max) IV on day 1 or each 21 day cycle for 6 cycles or until progression or unacceptable toxicity.

SUMMARY:
The purpose of this study is to evaluate whether treatment with a new drug called ZK-Epothilone (ZK-Epo) given with prednisone in patients with androgen-independent prostate cancer, who have not had previous chemotherapy, is safe and helps to decrease PSA (Prostate-specific antigen) levels.

DETAILED DESCRIPTION:
This study has previously been posted by Berlex, Inc. and Schering AG, Germany.Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc., Schering AG Germany has been renamed to Bayer Schering Pharma AG, Germany. Bayer HealthCare Pharmaceuticals, Inc.and Bayer Schering Pharma AG, Germany are the sponsors of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Must have evidence of confirmed metastatic prostate cancer
* Serum testosterone must be less than 50 ng/mL
* Disease must be progressing despite anti-androgen therapy
* PSA level must be elevated
* Additional criteria determined at screening visit

Exclusion Criteria:

* Any previous cytotoxic chemotherapy for prostate cancer
* Use of any investigational drug in the last 4 weeks
* Symptomatic brain tumors requiring radiation to the brain
* Active infection
* Additional criteria determined at screening visit

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-08-01 (Actual); Primary Completion 2008-09-24 (Actual); Study Completion 2009-12-21 (Actual)

PRIMARY OUTCOMES:
PSA Response to treatment with ZK-Epo plus prednisone after 6 cycles | at least 28 days post day 21 of last cycle of treatment

SECONDARY OUTCOMES:
Safety & Tolerability of ZK-Epo plus prednisone | until progression, unknown duration

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (15):
- United States (12):
  - Fountain Valley, California
  - Sarasota, Florida
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - Billings, Montana
  - Omaha, Nebraska
  - The Bronx, New York
  - Canton, Ohio
  - Portland, Oregon
  - Altoona, Pennsylvania
  - Fort Worth, Texas
  - Seattle, Washington
- Argentina (3):
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Buenos Aires
  - Córdoba

REFERENCES:
- [Result] Beer TM, Smith DC, Hussain A, Alonso M, Wang J, Giurescu M, Roth K, Wang Y. Phase II study of first-line sagopilone plus prednisone in patients with castration-resistant prostate cancer: a phase II study of the Department of Defense Prostate Cancer Clinical Trials Consortium. Br J Cancer. 2012 Aug 21;107(5):808-13. doi: 10.1038/bjc.2012.339. Epub 2012 Jul 31. PMID 22850553